CLINICAL TRIAL: NCT06359769
Title: Group Cognitive Evolutionary Therapy for Depression - A Randomized Clinical Trial
Brief Title: Group Cognitive Evolutionary Therapy for Depression
Acronym: GRCET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bucharest (Other)
Responsible Party: Principal Investigator, Cezar Giosan, Associate Professor of Psychology, University of Bucharest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GROUPCET
Record Dates: First submitted 2024-04-06; First posted 2024-04-11 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Depression; Anxiety
Keywords: Evolutionary Psychology; Evolutionary Psychopathology; Group Therapy; Cognitive Behavioral Therapy; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Cognitive Evolutionary Therapy (Experimental): In-person therapy groups
  Interventions: Behavioral: Group Cognitive Evolutionary Therapy
- Waitlist (No Intervention): Waitlist. No intervention for this arm.

INTERVENTIONS:
Behavioral: Group Cognitive Evolutionary Therapy — In-person therapy group. Delivery method: in-person groups. Number of sessions: 2. Duration of each session: 8 hours. Topics to be covered in the sessions are informed by the answers to the Fitness Evaluation Scale, following an adapted protocol of Cognitive Therapy for Depression.
  Arms: Group Cognitive Evolutionary Therapy

SUMMARY:
The goal of this clinical trial is to measure the effects of Group Cognitive Evolutionary Therapy on mental health, especially on depressive symptoms and anxiety.

Participants will be allocated in one of two conditions: (1) Group Cognitive Evolutionary Therapy (intervention) or (2) Waitlist. The intervention will consist of two 8-hour sessions of Group Cognitive Therapy, in two consecutive days.

The Group Cognitive Evolutionary Therapy group will be compared to the waitlist group to test the efficacy of the intervention.

DETAILED DESCRIPTION:
The aim of the study is to assess the efficacy of Group Cognitive Evolutionary Therapy on depressive symptoms and other indicators of mental health for people with mild to severe depressive symptoms. This clinical trial will provide essential insights into the potential benefits of this form of therapy. The results will contribute to the development of a short, economical and effective method of enhancing mental health for patients with mild to severe depressive symptoms.

After recruitment, participants will be randomly assigned to one of two conditions: (1) Group Cognitive Evolutionary Therapy (intervention) or (2) Waitlist.

The intervention group will participate in two 8-hour sessions of Cognitive Evolutionary Therapy over two consecutive days, in groups of no less than 5 and no larger than 8 people. These groups will be led by licensed psychologists with extensive knowledge of evolutionary psychology and cognitive evolutionary therapies.

Both groups will be evaluated at (1) pre-intervention (baseline), (2) one week after the intervention, and (3) three months after the intervention.

G*Power analysis yields a total of N = 44 (f = 0.25, power = 0.95) for the two conditions.

The statistical analysis plan includes the analysis of primary and secondary outcomes, which will be assessed using predefined measures described at the measures section. Additionally, the investigators will assess various predictors to gain insights into the factors influencing intervention outcomes. These predictors will be measured using specific instruments, including screeners (Diagnostic and Statistical Manual, Fifth Edition - Text Revision Self-Rated Level 1 Cross-Cutting Symptom Measure-adult version and The Personality Inventory for Diagnostic and Statistical Manual, Fifth Edition-Brief Form-adult version), and the Adverse Childhood Experiences questionnaire to assess adverse childhood experiences.

Besides demographic assessors and the above mentioned instruments, The Evolutionary Fitness Scale will be used both to determine predictors for the intervention outcome and as an assessment tool for the topics of interventions for each subject, this being a central part of Cognitive Evolutionary Therapy.

ELIGIBILITY:
Inclusion Criteria:

* mild to severe depressive symptoms
* age 18 to 65

Exclusion Criteria:

* severe personality traits (antagonism, impulsivity, disinhibition, psychoticism)
* formally diagnosed with a severe mental disorder
* currently participating in any ongoing therapeutic intervention for mental health.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Depressive symptomatology | up to 6 months
  Depressive symptomatology will be assessed with the 21-item Depression Anxiety and Stress Scale (DASS 21). Participants assign ratings on a scale of 0 to 3 based on how often they experienced specific items in the preceding 1-week timeframe (0- not at all; 3 - nearly every day). The depression subscale is a 7-question self-reported instrument that assesses dysphoria, hopelessness, devaluation of life, self-depreciation, lack of interest, anhedonia and inertia. Clinical cutoffs are provided.
Anxiety symptomatology | up to 6 months
  Anxiety symptomatology will be assessed with the Depression Anxiety and Stress Scale (DASS 21), a set of three self-report scales designed to measure the emotional states of depression, anxiety, and stress.
  The anxiety scale is a 7-question self-reported instrument designed to assess autonomic arousal, skeletal muscle effects, situation, anxiety, and subjective experience of anxious affect. Participants assign ratings on a scale of 0 to 3 based on how often they experienced specific items in the preceding 1-week timeframe (0 - not at all; 3 - most of the time). The total score for the seven items ranges from 0 to 21 and is a dimensional value.

SECONDARY OUTCOMES:
Sleep quality | up to 6 months
  Sleep quality will be assessed with a single item Sleep Quality Scale (SQS). Participants rate their overall sleep quality for the majority of nights in the past seven days on scale from 0 to 10, (0 - terrible, 10 - excellent)
Stress | up to 6 months
  By employing the Depression Anxiety and Stress Scale (DASS 21) stress will be measured by the stress subscale, sensitive to chronic non-specific arousal. The stress subscale measures difficulty relaxing, nervous arousal and being easily upset, agitation, irritability, over-reactivity, and impatience.
Social provisions | up to 6 months
  Social provisions will be assessed with the 10-item Social Provisions Scale (SPS 10). Each of the 10 questions will be answered on a scale from 1 to 4 (1- strongly disagree, 4 - strongly agree) with reference to the current relationship with friends, family members, coworkers, community members and others.
Satisfaction with life | up to 6 months
  Satisfaction with life will be measured with the Satisfaction With Life Scale (SWLS). The scale consists of 5 items designed to measure global cognitive judgments of one's life satisfaction. Participants indicate how much they agree, or disagree with each of these 5 items using a 7-point scale that ranges from 1 (strongly disagree) to 7 (strongly disagree).
Self-perceived mate value | up to 6 months
  Each subject's self perceived mate value will be measured with the Components of Mate Value Survey (CMVS). The survey consists of 22 questions with reference to various dimensions of self perceived mate value, and can be answered on a scale from 1 to 5 (1 - strongly disagree, 5 - strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Cezar Giosan, PhD, Study Chair — University of Bucharest
Locations (1):
- University of Bucharest, Bucharest, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giosan, C. (2020). Cognitive Evolutionary Therapy for Depression. Springer International Publishing. https://doi.org/10.1007/978-3-030-38874-4.